CLINICAL TRIAL: NCT04262453
Title: Obstructive Sleep Apnea Syndrome In Patients Treated For Cancer Of The Upper Aerodigestive Tract : The SAOS-K Study
Brief Title: Obstructive Sleep Apnea Syndrome In Patients Treated For Cancer Of The Upper Aerodigestive Tract
Acronym: SAOS-K
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A02373-52
Record Dates: First submitted 2019-12-09; First posted 2020-02-10 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Upper Aerodigestive Tract Neoplasms; Obstructive Sleep Apnea-hypopnea Syndrome
Keywords: Upper Aerodigestive Tract Neoplasms; Obstructive Sleep Apnea-hypopnea Syndrome; Epworth score; Ventilatory Polygraphy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective open-label, non-randomized, monocentric, cohort study, to assess the prevalence and severity of sleep apnea syndrome in patients treated for cancer of the upper aerodigestive tract.

The patient follows a usual course of care including, at the end of the treatment of his cancer of the upper aerodigestive tract, screening for obstructive sleep apnea syndrome at 3 months and 6 months (Epworth score and ventilatory polygraphy)

DETAILED DESCRIPTION:
Prospective open-label, non-randomized, monocentric, cohort study, to assess the prevalence and severity of sleep apnea syndrome in patients treated for cancer of the upper aerodigestive tract.

Patients are included in the study when they are hospitalized for panendoscopy. Thereafter, it takes about 1 month to start any treatment. The duration of treatment is estimated at about 5 months (the longest regimen would be induction chemotherapy followed by surgery and adjuvant complementary treatment). After which the patient follows a usual course of care including, at the end of the treatment of his cancer of the upper aerodigestive tract, screening for obstructive sleep apnea syndrome at 3 months and 6 months (Epworth score and ventilatory polygraphy).

ELIGIBILITY:
Inclusion Criteria:

* macroscopic lesion suggestive of a cancerous tumour of the upper aerodigestive tract (oral cavity, oropharynx, larynx, hypopharynx, cavum, cervical lymph node metastases with an occult primary cancer)
* awaiting anatomopathological confirmation

Exclusion Criteria:

* history of cancer of the upper aerodigestive tract
* history of known obstructive sleep apnea syndrome
* cancer of the thyroid, salivary glands, nose and paranasal sinuses
* patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a recently discovered upper aerodigestive tract tumour who have not yet started treatment
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Occurence of obstructive sleep apnea syndrome | 3 months after the end of treatment for cancer of the upper aerodigestive tract
  Obstructive sleep apnea syndrome is defined by an apnea-hypopnea index greater than or equal to 15 per hour

SECONDARY OUTCOMES:
Delay in onset of obstructive sleep apnea syndrome after completion of cancer treatment | during the 6 months follow-up
  Delay in onset of obstructive sleep apnea syndrome after completion of cancer treatment
Epworth score | at 3 months and 6 months
  The Epworth auto-questionnaire, rated from 0 (better) to 24 (worse), assess day-time sleapiness.
Occurence of obstructive sleep apnea syndrome | 6 months after the end of treatment for cancer of the upper aerodigestive tract
  Obstructive sleep apnea syndrome is defined by an apnea-hypopnea index greater than or equal to 15 per hour

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Baron, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huyett P, Kim S, Johnson JT, Soose RJ. Obstructive sleep apnea in the irradiated head and neck cancer patient. Laryngoscope. 2017 Nov;127(11):2673-2677. doi: 10.1002/lary.26674. Epub 2017 May 23. PMID 28543072
- [Result] Gilat H, Shpitzer T, Guttman D, Soudry E, Feinmesser R, Bachar G. Obstructive sleep apnea after radial forearm free flap reconstruction of the oral tongue. Laryngoscope. 2013 Dec;123(12):3223-6. doi: 10.1002/lary.24125. Epub 2013 Apr 10. PMID 23575744
- [Result] Loth A, Michel J, Giorgi R, Santini L, Rey M, Elbaum JM, Roux N, Giovanni A, Dessi P, Fakhry N. Prevalence of obstructive sleep apnoea syndrome following oropharyngeal cancer treatment: A prospective cohort study. Clin Otolaryngol. 2017 Dec;42(6):1281-1288. doi: 10.1111/coa.12869. Epub 2017 Apr 18. PMID 28332763
- [Result] Faiz SA, Balachandran D, Hessel AC, Lei X, Beadle BM, William WN Jr, Bashoura L. Sleep-related breathing disorders in patients with tumors in the head and neck region. Oncologist. 2014 Nov;19(11):1200-6. doi: 10.1634/theoncologist.2014-0176. Epub 2014 Oct 1. PMID 25273079